CLINICAL TRIAL: NCT04626661
Title: Mitochondrial Oxygen Measurement Variability in Critically Ill Patients: Validation of the COMET Measurement System
Brief Title: Mitochondrial Oxygen Measurement Variability in Critically Ill Patients (INOX Variability Study)
Status: Completed | Type: Observational
Sponsor: Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.G. van der Bom, Professor J.G. van der Bom, Sanquin-LUMC J.J van Rood Center for Clinical Transfusion Research
Other Study IDs: NL71914.058.19
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Mitochondrial Oxygenation Measurement; Measurement Error; Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health volunteers: The study population will consist, initially, of healthy volunteers. This group was chosen to perform measurements on, to eliminate the effect of critical illness and interventions on the critically ill patients and to better explore the effect of time-since-application of the 5-aminolevulinic acid-patches.
  Interventions: Device: COMET measurement system
- Patients admitted to the ICU after neurosurgery: This study population will consist of patients undergoing elective neurosurgery with planned postoperative recovery of at least 24 hours in the intensive care unit or medium care unit. Leiden University Medical Center is a neurosurgical center in which a wide variety of surgeries including tumor resection in the posterior cranial fossa (including vestibular schwannoma) are performed. Clinical experience has shown that this cohort of patients are in general, hemodynamically the most stable patients and receive the least amount of interventions compared to other cohorts of patients in the intensive care unit and medium care unit. For these reasons, the cohort of elective neurosurgical patients would be ideal to investigate the reason of the increased between- and within-subject variability of mitochondrial oxygen tension in the intensive care unit and medium care unit setting.
  Interventions: Device: COMET measurement system

INTERVENTIONS:
Device: COMET measurement system — Photonics Healthcare B.V. has developed an innovative non-invasive bedside monitoring system to measure Cellular Oxygen METabolism (the COMET).The COMET's non-invasive cutaneous mitoPO2 measurements rely on the protoporphyrin IX-triple state lifetime technique (PpIX-TSLT). This technique measures oxygen by oxygen-dependent quenching of delayed fluorescence lifetime of 5-aminolevulinic acid-induced mitochondrial PpIX (protoporphyrin IX). PpIX is the final precursor of haem in the haem biosynthesis pathway and is synthetized in the mitochondria. Administration of exogenous 5-aminolevulinic acid enhances PpIX to detectable levels and enhances mitochondrial origin of the delayed fluorescence signal. Measurements are based on the detection of time of extinction of red light emitted by the tissue following excitation with green light. The technique has been tested and calibrated for use in isolated organs and in vivo.

SUMMARY:
To determine the between- and within-subject variability of the mitochondrial oxygenation measurement with the COMET device over time in healthy subjects and in hemodynamically stable subjects admitted to the intensive care unit.

DETAILED DESCRIPTION:
Rationale:

Recent studies have shown the potential of a protoporphyrin IX-triple state lifetime technique to measure mitochondrial oxygen tension (mitoPO2) in vivo, which possibly is an early indicator of oxygen disbalance in the cell. With the advent of the COMET measurement system, steps have been made to determine the feasibility of this measurement method. The INOX ICU-2 study (parent study) aims to tailor transfusion therapies to individual intensive care unit (ICU) patients based on mitochondrial oxygen tension. In the pilot study of the INOX ICU-2 study, in which the COMET measurement system was used on critically ill patients receiving red blood cell transfusion, an increase in the between- and within-subject variability was observed over time. This deviation was not explored during the development of the COMET measurement system. Therefore, we aim to determine the between- and within-subject variability of this measurement in healthy subjects and in hemodynamically stable subjects at the intensive care unit.

Main objectives:

To describe the between- and within-subject variability of mitoPO2 measurements during a 24 hour period after 5- aminolevulinic acid (ALA)-induction among healthy volunteers and among neurosurgical patients admitted postoperatively to the ICU or MC. Healthy subjects allow for the exploration of the effect of time-since-application of ALA-patch and neurosurgical patients allow for the exploration of a possible effect of ICU-admittance.

Study design:

Prospective cohort study.

Study population:

Healthy volunteers and neurosurgical patients admitted at the ICU or Medium Care(MC) of LUMC after surgery.

Study procedure:

MitoPO2 measurements will be taken in healthy volunteers using two ALA-patches offset to each other by 3 hours, this has been done to observe possible differences in measurements at different time-points after ALA-induction while maintaining other variables stable. Following the healthy volunteers, neurosurgical patients will be included. Patients will undergo neurosurgery as planned and common practice is that no major interventions are needed in the postoperative phase on the ICU/MC. At multiple predefined moments after surgery, mitoPO2 measurements will take place, again using two ALA-patches with a 3 hour offset.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The risks are small in this study with no serious adverse events (SAE) known. The burden for participants is small since it involves a non-invasive measurement. We will perform this study first in health volunteers. Following the healthy volunteers, neurosurgical patients will be included. Patients will undergo neurosurgery as planned and common practice is that no major interventions are needed in the postoperative phase on the ICU. Normal clinical practice will continue and will not be altered. These patients will allow for the exploration of a possible effect of ICU admittance.

ELIGIBILITY:
Inclusion Criteria:

* Age of patient is at least 18 years
* Healthy participants, defined as the absence of active or chronic disease (applicable only to healthy volunteer group).
* Patients are admitted to the ICU or MC after neurosurgery (applicable only to neurosurgery group).

Exclusion Criteria:

* patients without a legal representative in case the patient is not able to give informed consent
* pregnant or breast feeding women since there is no adequate data from the use of ALA in pregnant or breast feeding women
* patients with porphyria and/or known photodermatosis
* patients with hypersensitivity to the active substance or to the plaster material of ALA
* insufficient comprehensibility of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist, initially, of healthy volunteers. This group was chosen to perform measurements on, to eliminate the effect of critical illness and interventions on the ICU and to better explore the effect of time-since-application of the ALA-patches. Neurosurgical ICU/MC patients will subsequently be included to further explore the effect of critical illness (ICU admission). Since this cohort of patients receives minimal interventions, they are ideal to limit potential affecters on the between- and therefore also the within-subject variability.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Within-subject variability of mitochondrial oxygenation measurements over a period of 24 hours after ALA-induction | 24 hours
  To describe the between- and within-subject variability (assessed by standard deviation) of mitoPO2 measurements over a period of 24 hours after ALA-induction in healthy volunteers and in neurosurgical patients

SECONDARY OUTCOMES:
Between- and within-subject variability between 3 hour offset 5-aminolevulinic acid-patches | 24 hour
  The goal is to describe the difference in the between-subject and within-subject variability between 3 hour offset 5-aminolevulinic acid patches at each time point. The hypothesis is that seen differences can be attributed to the patches itself.
Safety of mitochondrial oxygenation measurements | 48 hours
  Description of the adverse and serious adverse events during and after mitochondrial oxygenation measurements, both in neurosurgical patients admitted to the intensive care unit or medium care unit after their operation, and in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: J. G. van der Bom, PhD, MD, Principal Investigator — Leiden University Medical Center; M. S. Arbous, PhD,MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baysan M, Broere M, Wille ME, Bergsma JE, Mik EG, Juffermans NP, Tsonaka R, van der Bom JG, Arbous SM. Description of mitochondrial oxygen tension and its variability in healthy volunteers. PLoS One. 2024 Jun 3;19(6):e0300602. doi: 10.1371/journal.pone.0300602. eCollection 2024. PMID 38829894